### Prospective Randomized Controlled Trial Comparing Resident Performance and Clinical Outcomes with Two Different Polypropylene Meshes for Laparoscopic Inguinal Hernia

#### NCT01825187

Study Protocol and Analysis Plan

Document Date: February 8, 2013

# New Hanover Regional Medical Center Institutional Review Board (IRB)

2131 South 17th Street/P.O. Box 9000 Wilmington, NC 28402-9000

| | PCE | ARCH | τΛ | וכוכו | 10 | Λ "T" 1 / | <b>∼</b> 8 | . 1 |
|---|------|------|-----|-------|------|-----------|------------|-----|
| П | (ヒンド | ARC | 1 A | PPI | 10:7 | 4 I II | ( ) r | V |

Consent Form Version Date:

| NHRMC: IRB ID# □Full Board □Expedited Review Cat | egory |
|---|---|
| Check the appropriate boxes to indicate the documents you are submitting. IRB Application (required for all studies) Informed Consent Protocol Recruitment Materials Dated/Current CV for PI only (if not currently on file in IRB office) Professional License/Certifications (if required for study) Data Collection Tool (QOL, CRF, Surveys, etc.) Other (i.e. Investigator Brochure) Administrative Attachment (required, one copy for Clinical Research Officer) Human Participant Protection Certificate (required all study staff if not currently on file in IRB office) Currently on file in IRB office) Submit application package double-sided & collated: Full Board: Original plus of the polications must "stand all should provide all information requested, i.e., complete and should provide all information answered directly on the form you may reference other documents with supporting information, or respond solely by stating "see attached". | copied 13 copies nal Only ne" and swers must ion. be m. While cuments do not |
| You must have administrative approval from the Clinical Research Officer prior to submission to the IF | lB as |
| evidenced by a signature below. To be completed by the Clinical Research Officer. | |
| Administrative Review Complete | |
| ☐ Administrative Approval Pending Clinical Research Officer Dat | е |

### Part I: Study Identification & Information

Version Date:

Complete the following information as it applies to your study.

Study Title Prospective Randomized Controlled Trial Comparing Resident Performance and Clinical Outcomes with Two Different Polypropylene Meshes for Laparoscopic Inguinal Hernias

Study ID Protocol Number: Amendment Date (if applicable):

| | Principal Investigator | Primary Study Coordinator |
|------------------|-------------------------|---------------------------|
| Name w/ Degrees | William Hope, MD | Chiquta Harris, BS |
| Practice/Company | SEAHEC Surgery | SEAHEC Research |
| Address | 2131 S 17th St | 2511 Delaney Ave. |
| City, State, Zip | Wilmington NC 28401 | Wilmington, NC 28403 |
| Phone | 910.667.9233 | 910.667.9253 |
| Fax | 910.763.4630 | 910.667.9343 |
| Pager | 910.341.5342 | |
| E-mail | William.Hope@SEAHEC.net | Chiquta.Harris@seahec.net |

# A. Investigator Research Experience

Version Date: 3/11

### NHRMC IRB

| | | | | Contraction Contra |
|---|---|---|---|---|
| ٦. | Has the PI ever conducted research | ☐ No | 🛛 Yes | Currently have an open study(ies). |
| | at NHRMC before? | Role: | | Participated within last 2 years. |
| | - Level - Leve | ⊠ PI | Co-Pl | Greater than 2 years. |
| 2. | Has any IRB ever taken corrective | ⊠ No | ☐ Yes | If yes, why? |
| | action for non-compliance including but not limited to issuance of a non- | | | |
| | compliant closure of any of the Pl's | | | |
| | studies? | | | |
| 3. | Is any special or technical training | ⊠ No | Yes | If yes, explain. |
| | required specific to the conduct of | | | |
| | the study? | | | |
| 4. | Name of course PI took for Human | l | | IH PHRP Cert. #129665 |
| <u> </u> | Participant Protection Education. | | | 11/05/2008 Expiration date: |
| 5. | Name of course Study Coordinator | l ' - ' | or course: Nate: | IH PHRP Cert. #819035 Expiration date: NA |
| | took for Human Participant Protection Education. | Comple | mon Dale. | Expiration date. 1470 |
| *N( | OTE: If you have not completed a cours | e in hum: | an particip | ant protections, there is a link on the IRB |
| we | bpage or go to http://phrp.nihtraining.c | om for a | n online tu | orial course. If you have completed a course |
| oth | ner than the NIH course, you will be requ | ired to pr | ovide a ca | py of the syllabus for the course. |
| В. | Nursing Research | | | |
| Co | omplete this section <b>only if the PI or C</b> | o-Pls are | e nurses. | ☐ This section is not applicable to my study |
| 1. | • | | · · = | es No PI |
| | Research Committee intra-hospital wel | | | es No Co-Pl |
| 2. | My contact information may be given | to the | = | es No Pl es No Co-Pl |
| | Nursing Research Committee to be listed | | | es No Co-Pl |
| | intra-hospital webpage as a resource t<br>nursing researchers. | O OII IEI | | |
| | Troising researchers. | | | |
| $\mathbf{c}$ | Investigational Agent | | | |
| | t investigational drugs/devices that o | are <b>not</b> E | DA appro | ved. |
| L13 | investigational arags, acrices that e | c <u></u> | 37. Gpp. 0 | This section is not applicable to my study |
| | Device *Complete section D belo | w | | Drug |
| No | ame: | | Gen | eric Name: |
| | 44-11-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1 | | | Prand Namo: |
| Mo | odel #: | | Bran | Brand Name: |
| IDI | E#: | | IND# | IND#: |
| L | Landers and the state of the st | | | |
| B. B I I I I I I I I I I I I | | | | |
| | Research Involving Devices | | انجامید | thath EDA and non EDA anniqued |
| Co | (both FDA and non-FDA approved). | | | |
| - | 140 | | Eval- | in. Devices are stored in the Operation Room |
| Where will the devices be stored? | | | | and are in stock in the OR holding room at New |
| | | | , , , | ver Regional Medical Center. |
| 2 | Who will receive and manage inventor | v for the | | e: OR Staff |
| devices throughout the study? | | | I ' ' | Nurses and Doctors |
| 3. | Who will have access to the devices? | | Nam | e: OR Staff |
| | | | | Title: Nurses and Doctors |
| 4. | How will the devices be accounted for | ś | | in. Devices that are availble on stock at the |
| | | | hosp | tal will be used and the Lot number will be |

recorded.

| 5. What protections are i improper use? | n place to prevent loss or | Explain. These are devices are currently FDA approved and used on a daily basis at NHRMC so there are already precautions in place to protect them. |
|---|---|---|
| Part II: Study Subjects and Procedures Complete the sections that apply to your study. A. Subject Enrollment and Demographics: This is a listing of the target study population. Check all that may apply. You don't have to meet the anticipated subject enrollment number, but you can't exceed it without an amendment to | | |
| increase the number an | | |
| ☐ Healthy Volunteers | Chronically III | Placebo (non active medicine) |
| Employees | Mentally III | ☐ No Treatment Condition (control group is |
| Students | Terminally III | involved that receives no study-related |
| ☐ Hospitalized Patients | Use of Banked Specimer | ns treatment) |
| Male Male | Use of Fetus/Fetal Tissue | Storage of Specimens for Future Use |
| | ★Indigent/Uninsured | Multi-center Study: Subject Enrollment |
| ■ Adults | ×Non-English Speaking | anticipated subject enrollment |
| Children (under 18) | ★Limited or No Literacy | # anticipated this site |
| (complete section V) | | Single Site Study: Subject Enrollment |
| *Pregnant (see below) | | # anticipated this site 511 |
| *The subject population | is in bold font represent pro | tected populations. If you are excluding subjects |
| because they are preg | nant, indigent/uninsured, n | on-English speaking, or limited or no literacy |
| please explain why: Pre | eanant women are exclude | ed from the study because they are not usually |
| operated on until after | | , |
| | They have delivered. | |
| B. Research Involving Children Complete this section only if study subjects are less than 18 years of age. Special requirements: 45 CFR 46 Subpart D – Additional Protections for Children Involved as Subjects in Research This section is not applicable to my study | | |
| Age of Pediatric Subject Preterm Newborn | cts (check all that apply) | |
| Term Newborn Inf | | |
| | Infants and Toddlers (28 days to 23 months) | |
| Children (2—11 years) Adolescents (12—18 years) | | |
| Special Protections (an | Special Protections (answer as applicable to your study) | |
| 1. Yes No | Does the research have a<br>subjects? Explain: | an identifiable prospect of direct benefit to the |
| 2. Tes No | | ieved through alternative means? Explain: |
| 3. Yes No No | N/A If using a placebo contro<br>Explain: | ol, does this place the subject at greater risk? |
| 4. Yes No N | V/A Will permission be sought | from both parents? If not, why? |
| 5. Yes No 6. Yes No | • | who are wards of the state? Explain: hat call for the presence of an advocate during |

# **Research Application**

| | consent proce | dures? If s | o, what? | Who? |
|---|---|---|---|---|
| 7. | | | | conduct of the research? If not, why? |
| 8. | ☐ Yes ☐ No ☐ N/A Are mechanism | ns in place | to ensure | the child's dignity is not undermined |
| 0 | | | | ssent, etc.)? Explain:<br>eeds of adolescents (protection of |
| 9. | | | | ces, drugs, alcohol, etc.}, counseling, |
| | appropriate re | | | |
| 10. | How will parental permission be obtained | | □ N/A | Explain if applicable. |
| 11. | How will assent be obtained? This is gene | | □ N/A | Explain if applicable. |
| | written consent for children who can rea | | | |
| | -17. A script can be used for children unverbal permission. <b>Attach copies to your</b> | der / for | | |
| | submission. | | | |
| 12. | For research involving children under 8 years | ears of | □ N/A | Explain if applicable. |
| | age, what non-verbal cues will you watc | | | |
| | indicate the child is ready to end or paus<br>participation? | е | | |
| | рапсравон | | 1 | 4400 |
| C. | Confidentiality and Informed Cons | sent: Be s | pecific to | protections that will be in place for |
| | ojects. | | | |
| 1. | Where is study subject data kept? Check | : all that | │ □ Spc | onsor's Location |
| | apply. | | ⊠ Me | dical Record |
| İ | | | ☑ Prin | icipal Investigator/Local Research Office |
| | | | Oth | ner |
| 2. | Will precautions be taken to protect | □ No | Yes | Explain. All records will be coded and kept in |
| | subject information (e.g. locked file | | | a locked file cabinet. No patient or resident |
| | cabinet, password protected files, etc.). | | | identifiers will appear on any coding sheets |
| | | | | or electronic databases. Electronic |
| | | | | databases will be password protected. Strict |
| | | | | confidentiality will be maintained and no |
| | | | | patient or resident will be identified in any |
| | | | | report of our findings. A master list of patients |
| | | | | and residents will be maintained separately |
| | | | | from the coding sheets and databases. |
| 3. | Will the subject's personal health | ⊠ No | Yes | If yes, explain. |
| | information be released with identifiers | | | |
| | such as name, DOB, SSN? | | | |

| 4. | Are you requesting a waiver of consent? | No Yes | If yes, explain. A waiver of written consent is |
|---|---|---|---|
| | If no, complete questions 5-12. Waiver | | being requested for the residents involved in |
| | can only be requested if it makes your | | the study because the research presents no |
| | study infeasible to conduct. Answer "No" | | more than minimal risk of harm to subjects |
| | and indicate in the explanation if you | | and involves no procedures for which written |
| | plan to use implied consent language for | | consent is normally required outside of the |
| | a survey, or a telephone consent script. | | research context. The normal consenting |
| | | | process will apply to the patients. |
| 5. | Who will obtain informed consent? Only | Name and crede | entials: William Hope, MD |
| | the PI or Co-PIs may obtain consent. Refer | Study Role (PI / C | o-PI): PI |
| | to NHRMC policy on informed consent. | | |

| 6. | Describe how and where informed | If the subject is a p | potential candidate for the study, the subject |
|---|---|---|---|
| | consent will be obtained? | will be approache | ed by Dr. Hope. Dr. Hope will explain the study |
| | | to the subject. If the subject decides to participate in the study, he/she will be given the informed consent document to review | |
| | | and sign. Once ve | erbal consent is received, Dr. Hope will obtain |
| | | _ | om the subject. All documents will be written |
| | | | in a language to be understood by the |
| | | • | al time to review the informed consent |
| | | - | provided if needed. Consent will be obtained |
| | | | g the patient's pre-operative appointment or |
| | | • | NHRMC. Patients will be consented by Dr. |
| | | J | atient Surgery Clinic, SEAHEC Physicians' |
| | | · · | lurgical Units at NHRMC and/or the |
| | | • • | rtment. Dr. Hope will review the surgical |
| | | procedure and all of the steps associated with participating in | |
| | | the study. Dr. Hope will also review the informed consent | |
| | | documents with the patients. Patients will have a chance to ask | |
| | | Dr. Hope any questions they may have about the surgery and the study. Resident will be approached by Dr. Hope prior to the initiation | |
| | | | ope will give the residents the information |
| | | • | plain the study to the residents. Additional time |
| | | to review the information sheet will be provided if needed. Dr. Hope will address and answer all concerns and questions of the | |
| | | residents pertaining to the study. If the residents agree to | |
| | | participate in the study, the study coordinator will obtain verbal | |
| | | consent from the consenting residents. The will be no repercussions to any residents that objects to being in the study. | |
| | | · | |
| | • | Will there be an opportunity for potential subjects to take the | |
| | | informed consent form home to consider the options and to | |
| | | | ion with family members? No X Yes |
| | - | If no explain why: | |
| 7. | , | □ No ⊠ Yes | Explain. If necessary, a Spanish interpreter |
| | subjects, will the consent form be in their | □ N/A | will be used to explain the study and consent |
| | native language? If not, explain the | | process. |
| | process for consent. | | |

# **Research Application**

| 8. | If the subject is unable to provide | | ⊠ No | | Yes | If yes, explain. |
|---|---|---|---|---|---|---|
| | consent, will consent be obtained from | ı a | | | | |
| | legally authorized representative? | | | | | |
| 9. | If yes to Q.7, if the subject becomes ab | ole | ☐ No | | Yes | If no, explain. |
| | to provide consent, will you re-consent | ś | $\boxtimes$ | N/A | ` | |
| 10. | How will you ensure that only the | | Explain. Study consent and information sheets will only be | | | |
| | approved and current consent form is | i | printed | l as r | need | ed and no additional copies will be printed. |
| | used (e.g. only approved version will b | e | Only th | e ap | oprov | ed version of the consent form and the |
| | available, will print original each time, | | informo | ation | shee | et will be provided to the patients and residents. |
| | etc.)? | | The mo | ost c | urren | electronic version of the consent and |
| | | | informa | ation | shee | et will be kept in a separate electronic folder |
| | | | from p | rior c | conse | nt forms and information sheets to avoid |
| | | | printing | g the | wro | ng version. All previous drafts will be deleted. |
| 11. | Where will the original signed and date | ed | Locatio | on: C | r. Ho | pe's Office and/or SEAHEC Research |
| | informed consent form be maintained | ś | Department | | | |
| | | | A signed copy will be given to the subject? | | | |
| | | | □ No ⊠ Yes □ N/A | | | |
| | | | A signe | ed c | ору ч | vill be maintained in subject's medical record? |
| | | | □ No ⊠ Yes □ N/A If no, explain. | | | |
| 12. | Will the informed consent process be | | ☐ No | $\boxtimes$ | Yes | Explain. The informed consent process will be |
| | documented in the subject's medical | | | ] N// | A | documented in the subjects' medical |
| | record? (e.g. documented discussion | of | | | | records. There will be documentation of the |
| | risks/benefits, alternatives to study | | | | | discussion of the risks/ benefits associated |
| | participation, voluntary participation o | and | | | | with the study, any questions the subject had |
| | measures of understanding) | | | | | about the study, whether or not the subject |
| | | | | | | chose to participate in the study, and |
| | | | | | | evidence that the subject has a solid |
| | | | | | | understanding of what participation in the |
| | | | | | | study entails. |
| | | | ! | | | |
| | Recruitment: Tell how prospective | | | <u>ill be</u><br>Ye | | |
| 1. | Is there any prior relationship with | <b>⊠</b> 1 | NO 12 | א ופ | | f yes, explain. Patients may be current and/or |
| | the subjects and the PI? (one or | | | | ı | previous patients of the investigator. Dr. Hope |
| | both may be checked as | | | | | serves as the assistant professor to surgical |
| | applicable) | | | | | esidents. |

# **Research Application**

| 2. | If you as the PI are a clinician, will | | No | $\boxtimes$ | Yes | If no, explain how subjects will be identified. |
|---|---|---|---|---|---|---|
| | subjects be drawn exclusively from | | | | | |
| | your own sample base? | | | | | |
| 3. | If no to Q2, will the subject's | | No | | Yes | If no, explain. |
| | physician be consulted, contacted, | | | | | |
| | or notified? | | | | | |
| 4. | Will recruitment materials be used | $\boxtimes$ | No | | Yes | If yes, what types, and when and how will they |
| | (videos, ads, flyers, etc.)? | | | | | be used? |
| 5. | Will subjects be paid for | $\boxtimes$ | No | | Yes | If yes, explain. |
| | participating in the study, including | | | | | |
| | but not limited to compensation for | | | | | |
| | time, travel, etc.? | | | | | |
| 6. | Describe how subjects will be initially o | cont | acted | l (i.e | . recru | itment materials, letter, office visit, etc.)? Subjects |
| | will be initially contacted by Dr. Hope | at t | heir pr | eop | erativ | e visit. |
| L | | | | | | |
| | Benefits: Do not list monetary pay | me | nts as | <u>a b</u> | enefi | t. |
| 1. | Are there benefits to the subject? | | Explai | n. In | iere ar | e no direct benefits to research participants. |
| | (What are the benefits, if any, to the | | | | | |
| | subject by participating in the study?) | 1 | | | | |
| 2. | Are there benefits to society? (What | | • | | | ormation gathered from the study may benefit |
| | potential benefits to future individuals | | | • | | indergoing hernia surgery by determining which |
| | may the study provide?) | | | | | or use during these procedures. The study will |
| | | - 1 | | | | dge on the different types of hernia meshes and |
| | | | the le | ngth | of tim | ne it takes residents to perform the procedure. |
| | | | | | 1 11. | |
| F. | Costs to Subjects: Explain the find routine care costs. | anc | iai liai | DIIII | / 10 IN | e study subject; distinguish study related costs |
| 1. | | | N | 0 | X Y | es Explain. Participants will be responsible for |
| | subjects that are not paid by the | | | | | covering routine care costs associated with |
| | study? | | | | | doctor visits and the surgery. However, there |
| 2. | Will the subject be financially | | X N | lo | Y | es are no extra costs associated with this study. |
| | responsible should insurance deny | | | | | The six (6) month and one (1) year follow-up |
| | coverage of study-related costs? | | | | | visit are not routine, therefore, the patient will |
| 3. | Will the subject be financially | | | lo | X Y | not be charged for any of these services |
| | responsible should insurance deny | | | | | (both clinic and professional fees will not be |
| | coverage of routine care costs? | | | | | billed to the patients). For the 6 month and 1 |

| NHRMC IRB | | | Research Application |
|---|---|---|---|
| 4. Will the PI or a representative discuss | ☐ No | | year follow-up the patient will be contacted |
| with the subject the difference | | | by telephone or be asked to return to the |
| between study related costs and | | | SEAHEC Physician's Office. Dr. Hope will |
| routine care costs, and that the subject | | | discuss this information with the |
| or the subject's insurance provider will | | | patients. |
| be responsible for routine care costs? | | | |
| G. Statistical Analysis | | | |
| Who will provide statistical analysis? | | SEAHEC | Research Department |
| 2. Is there a data safety monitoring board? | | ⊠ No | Yes |
| | | □ N/A. | this is not a clinical trial or treatment study |
| Part IV: Description of Proposed Research Study NOTE: This portion of the application is not intended for a cut and paste from the protocol, but rather for a summary of why the study is needed and how the study will work at this institution. Please use lay terms or provide definitions. | | | |
| 1. Purpose and rationale: Provide a brief summary of the background information to put the study in context, include references and prior research as appropriate. State the research question(s) and tell why the study is needed or important. Describe the primary objective and any secondary objectives. Document a clear, concise purpose statement. If the study is a clinical trial involving patients as subjects and use of placebo, please justify the use of these controls. | | | part of the lower intestine, bulges through a coint in the lower abdominal wall. The bulge curs from this hernia can be extremely painful es not go away on its own. Inguinal hernia one of the most common operations and by general surgeons in the world. There o main ways to repair an inguinal hernia, open roscopic. |

incision in the groin (the fold or hollow on either side of the front of the body where the thigh joins the abdomen) so it is possible for the surgeon to see the entire area and perform the surgery without the use of a laparoscope (an instrument through which structures within the abdomen and pelvis can be seen). Open repairs lead to more scarring and a longer recovery period. A laparoscopic repair is done by making a small cut in or just below the belly button. The abdomen is then inflated with air to allow the surgeon to be able to see all of the organs. Then, a lighted scope called a laparoscope is inserted into the incision so the surgeon can see inside the abdomen during the surgery. Surgical instruments used to repair the hernia are inserted through other small openings in the abdomen and a mesh is placed over the bulge (hernia) to reinforce the abdominal wall. Laparoscopic repair has become an accepted standard for inguinal hernia repair and has become the technique of choice for recurrent inguinal hernias.

One main part of the procedure to repair a hernia involves the placement of a prosthetic (a device that substitutes for missing parts or pieces) mesh to reinforce the abdominal wall and allow for a tension free repair. The use of the mesh also helps to lower the recurrence rate (the chance that the hernia will come back). The most common type of mesh prosthesis that is placed in laparoscopic inguinal hernias is a polypropylene (the substance the mesh is composed of) mesh which has been shown to be safe and effective.

There is some emerging evidence that a "lighter weight" form of this mesh may improve quality of life outcomes following surgery and is the mesh currently being used at New Hanover Regional Medical Center for laparoscopic inguinal hernia repair. However, there are many different "light weight" polypropylene meshes on the market that are FDA approved and available for use. Currently, there are two different forms of the mesh being used interchangeably for the procedure at NHRMC. Both of these meshes have had good clinical outcomes.

The purpose of this research study is to evaluate the clinical effectiveness of the two meshes currently being used. The study may provide evidence on whether one mesh is more effective than the other. A secondary goal of the study is to evaluate the ease of use and time it takes residents to place and perform the surgery using these two different meshes. This information may make it possible to determine if one mesh is easier for residents to use during surgery and therefore take them less time to perform the procedure.

The effectiveness of the meshes will be measured by the patient's length of hospital stay, perioperative complications, recurrence rate, patient pain score and/or comfort level and the patient's postoperative quality of life.

- Description of study design, methods, and procedures, describe the study in sequential order as it is to be conducted at this institution. The following should be included:
- > type of experimental design
- study procedures: a sequential description of what will be asked of/done to subjects (to include identification and recruitment of subjects, consent process, treatment or intervention if applicable, length of participation, additional visits, follow-up, etc.)
- description and assignments of subjects to various arms of the study (if applicable)

This will be a prospective open-label randomized study conducted by Dr. Hope from the study's approval date to until December 31, 2015. Approximately five-hundred (500) subjects will be enrolled in this study.

Patients presented to NHRMC, the Outpatient Surgery Clinic, SEAHEC Physicians' Office, Inpatient Surgical Units at NHRMC and/or the Emergency Department for abdominal wall hernia repair during their preoperative visit and who meet the inclusion and exclusion criteria will be counseled by Dr. Hope on surgical options for repair to determine if they would

- doses, frequency, and route of administration of medication and other treatment
- data that will be collected
- > primary outcome measurements
- follow-up procedures
- If the study involves clinical activities, distinguish routine care procedures from those that are study specific

rather undergo an open or laparoscopic repair. If the patient is a candidate and agrees with undergoing the laparoscopic repair, they will be asked if they would like to participate in a randomized trial comparing two different meshes. If the patient agrees, he/she will be presented with information regarding this study. The study will then be explained to the patient by Dr. Hope.

Dr. Hope will give the patients the informed consent document at New Hanover Regional Medical Center, Outpatient Surgery Clinic, SEAHEC Physicians' Office. Inpatient Surgical Units at NHRMC and/or the Emergency Department, Dr. Hope will review the page-by-page informed consent document with the patients. A copy of the informed consent document explaining the objectives and associated risks and benefits of the study will be given to the patient. The patient will be allowed to read and review the elements of the informed consent document. Patients will have a chance to ask Dr. Hope any questions they may have about the surgery and the study. If necessary, the patient will be allowed additional time to review the document. After receiving verbal consent, Dr. Hope will obtain written consent from the patient. A copy of the signed informed consent document will be given to the patient and another copy will be placed into the patient's medical record. The original document will be placed into a separate secure file cabinet that will be locked at all times.

On the day of surgery, patients agreeing to participate in the study will be randomized to receive either one of two meshes - ultrapro mesh (Ethicon) or bard 3d max (Bard). This randomization will occur with a random pattern being generated using an electronic random number generator. Then, the random assignments will be placed inside opaque, sequential envelopes. The envelopes will be opened, in order, which will guarantee a random assignment of subjects to each study arm.

Prior to the surgery, patients will be given the Carolinas Comfort Scale (CCS) and Visual Analog Scale (VAS). These study specific scales will be used to access the patients' pain and/or comfort level prior to surgery and should take no longer than 5 minutes to complete. The CCS uses a patient questionnaire of 8 questions to establish a quality measure for pain. Patients are asked to rate, on a scale of 0 to 5, sensation of mesh, pain and movement limitations during the following activities: lying down, sitting up, activities of daily living, coughing or deep breathing, walking or standing, walking up or down stairs, and while performing non-work related exercising. The VAS

helps patients to say how good or bad their health state is. This scale uses a line with two different extremes. The extremes can vary in forms. Some VAS can ask the patient to range their pain level or current health status on a rating of either 0-10 (with 0 being no pain and 10 being the worst possible pain) or by choosing a picture of a happy or sad face.

Patients with bilateral inguinal hernias (an abnormal opening or defect that occurs on both sides of the groin), either found preoperatively or intra-operatively, will be treated as one hernia and will have the same mesh placed on both sides. Cases will be performed by one attending using his standard technique for laparoscopic inguinal hernia repair.

Data to be collected will include the patients' demographic information (age, sex, race), comorbidities (if present), smoking history, drinking history, medications, allergies and previous surgeries.

Operative data will include the following: type of anesthesia (all patients will undergo general), technique of laparoscopic access, type and side of hernia (direct or indirect), size of mesh used, type and number of tacks used to secure mesh, operative time, blood loss, urine output, and type and technique of closure.

Postoperative data will include: length of hospital stay, perioperative complications, recurrence rate, patient pain score and patient's postoperative quality of life. Further follow up data will include an assessment of the patient's recurrence rate, pain scale and quality of life during the patient's 1-2 weeks, 6 months, and 1 year follow-up. The patient will also be asked to rate their pain and/or comfort level by using the CCS and/or the VAS. During their 1-2 weeks visit, the patient will be informed of the 6 and 1 year follow-ups. For the six (6) month and one (1) year follow-up the patient will be contacted by telephone and/or be asked to return to the SEAHEC Physician's Office. The patient will not be charged for any of these services. Subjects will be tracked and identified with the use of the research record that will be set up in EPIC. Patients will be associated with the study and their surgery admission will be associated with the study for billing and coding compliance. In case the above system does not work, as a secondary system, patients will be tracked using an excel spreadsheet.

Resident will be approached by Dr. Hope prior to the initiation of the study. Dr. Hope will give the residents the information sheet and will explain the study to the

residents. Additional time to review the information sheet will be provided if needed. Dr. Hope will address and answer all concerns and questions of the residents pertaining to the study. If the residents agree to participate in the study, the study coordinator will obtain verbal consent from the consenting residents. The will be no repercussions to any residents that objects to being in the study.

Resident level (PGY level), participation in the case (percentage of resident involvement to be determined by attending physician), time to perform the three critical portions of the case (laparoscopic access and takedown of peritoneum, placement of mesh, closure of peritoneum, and closure) will all be documented. This is routinely done by the surgical residents.

Following the case, the resident will be given a performance scale (NASA-TLX) to grade his/her performance in conducting the surgery. This is not routinely done but is done for some surgical cases. The NASA-TLX is a publically available, multi-dimensional scale designed to obtain workload estimates from one or more operators while they are performing a task or immediately afterwards. It contains 6 scales that will ask the residents to rate their mental demand, physical demand, temporal demand, performance, effort and frustration on a scale of very low to very high. This will take the resident no more than three (3) minutes to complete. Once the resident has completed the scale, they will return the scale to Dr. Hope. Dr. Hope will then give the scales to the study coordinator who will keep all the scales in a locked and secure place at SEAHEC. The scale will be linked to the study patient by entering the study patient's study ID number on the scale. The residents do not routinely complete the NASA-TLX for all surgeries but for some they do. The requirement for the completion of the NASA-TLX by the surgical residents will be new and specific for this study.

Descriptive statistics will be performed and outcomes and resident performance will be compared based on resident level and type of mesh used. A p-value of <0.05 will be considered significant.

3. Description of risks and measures to minimize risks:

Do not insert "No Risk", at minimal every study has arisk of breach of confidentiality.

Include risk of:

- breach of confidentiality,
- known side effects of study medication, risk of pain, and/or physical injury,

This study has no additional health risks. The short and long physical risks associated with hernia repair of both meshes include very mild pain and awareness of mesh and/or stiffness in the groin respectively. However, these risks are similar to the risks seen in routine surgical hernia repairs.

### **NHRMC IRB**

| * * De. | psychosocial harm (emotional distress, embarrassment, , etc.), economic harm (loss of insurability), legal jeopardy (disclosure of illegal activity) scribe the measures taken to minimize each risk. | As an additional safety precaution, once the first one hundred (100) subjects have been entered into the study by the Pl, an interim analysis (analysis of data collected at a certain time during the study in order to detect any trends of adverse events or to see if the study has negative effects on the patient's safety) will be conducted by the statistician. Any negative trends or adverse events will be reported to the IRB by the study coordinator. Another interim analysis will be collected by the statistician after the first two hundred and fifty (250) subjects have been entered into the study. Any negative trends or adverse events will be reported to the IRB by the study coordinator. The possible side effects and complications of the surgery relate to the procedure itself and will not be related to the data collection. |
|---|---|---|
| | | A possible risk may be the loss of privacy and the confidentiality of patient information. Access to the database is protected by password and is only accessible to the study and research staff. Every effort will be made to protect the privacy of patient information in the database, but this cannot be guaranteed. |
| 4. | Inclusion/exclusion criteria: List required elements of potential subjects and those that preclude enrollment. (Exclusion criteria are not opposite of inclusion criteria, but rather elements within the already identified subject population that would be a cause for exclusion from the study.) | The inclusion criteria for patients in this study will include all of Dr. Hope's patients undergoing laparoscopic repair for the treatment of either single or bilateral inguinal hernias from the study's approval date to December 31, 2015. The inclusion criteria for residents in this study will include all surgery residents. The exclusion criteria for patients in this study will include patients requiring emergency surgery, pregnant patients and patients under 18 years of age. |
| | | There is no exclusion criteria for residents in this study. |
| _ | | |

### Part V: Financial Conflict of Interest

This section is to be completed for all financially sponsored studies.

Are you being paid to conduct this study? 

Yes 

No

If yes, complete questions below, if no skip to next section.

If financially sponsored indicate source:

| | | marking YES or NO if any of the financial interests or arrangements described below apply spouse, or dependent children. |
|---|---|---|
| | • | |
| Yes | No | Compensation for services (e.g. consulting fees or honoraria), or in-kind payments, other than from the Investigator's primary employer, in the prior calendar year or project over the next twelve months. |
| | | Royalty income or the right to receive future royalties under the patent license or copyright, |

| | where the research is directly related to the licensed technology or work. |
|---|---|
| | Equity interests (e.g. stocks, stock options or other ownership interests, including equity holdings where the value cannot readily be determined by reference to public prices). |
| | Intellectual property rights (e.g. patents, copyrights, and royalties from such rights). |
| | Gifts or funds available to the researcher from this sponsor beyond the current research project. |
| | Funding expected to significantly exceed the projected costs of conducting the current research project. |
| | Any other financial or personal interest which presents an actual or perceived conflict of interest. |
| If the response to any item is yes, please provide below a full description of the financial interest (including amount of compensation and other information related to compensation) and how the financial interest might affect or be affected by the proposed research. | |
| I certify that the above information is complete and accurate, in accordance with 21 CFR Part 54. Furthermore, if changes occur in my financial arrangements and interests, or those of my spouse or dependent children, during the course of this study, I am required to update this form. | |
| Principal Investigator (Printed Name) Signature Principal Investigator | |

### Agreement of the Principal Investigator

- I certify that I have reviewed the information in this document and it is correct and complete.
- I certify that each of the named study personnel has accepted his/her role in this study.
- I agree to a continuing exchange of information with the New Hanover Regional Medical Center's (NHRMC) Institutional Review Board (IRB) as required by NHRMC IRB Policy and Procedure and the FDA Regulations and Guidelines.
- I agree to conduct this study according to the Good Clinical Practice Guidelines and regulations (FDA).
- Under non-emergent conditions, I agree to obtain IRB approval before making any changes or additions to the project. I will provide progress reports as required.
- I agree to report promptly to the IRB all unanticipated problems or serious adverse events involving risk to human subjects.
- A signed and dated copy of the consent form will be given to each subject and the
  original will be retained in the study files. If the study involves NHRMC patients, I will be
  responsible for placing a copy of the signed consent in the patient's medical record.
- I will notify the IRB in the event the study closes.

- I agree to use the patient health information as specified in this research study application and to:
  - Only view and obtain the information necessary to complete the scope of this study.
  - Only release information as it is specified in an approved and signed informed consent form.
  - Store the collected information in a confidential manner.
  - Comply with the standards and regulations set forth by the Health Information Management Department to acquire and use the medical records.
  - Be responsible for the study staff listed in this application or required attachments and ensure that they will abide by the rules of confidentiality outlined above.

| | 2574 | WILLIAM HOPE | 1/24/,3 |
|-----------|------|--------------|---------|
| Signature | 7 / | Printed Name | Dafe ' |

NOTE: Your signature must be legible for submission to be accepted.